CLINICAL TRIAL: NCT04450550
Title: Electrical Vestibular Neve Stimulation(VeNS) in the Management of Parkinson's Disease
Brief Title: Electrical Vestibular Nerve Stimulation (VeNS) in the Management of Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurovalens Ltd. (Industry)
Collaborators: R D Gardi Medical College, Ujjain (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVSPD001
Record Dates: First submitted 2020-06-11; First posted 2020-06-29 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator)
  Interventions: Device: VeNS device
- Sham (Sham Comparator)
  Interventions: Device: Sham VeNS device

INTERVENTIONS:
Device: VeNS device — VeNS treatment
  Arms: Active
Device: Sham VeNS device — Sham treatment of VeNS
  Arms: Sham

SUMMARY:
Parkinson's disease burdens an increasing number of elderly populations in the country.

Parkinson disease is a chronic, progressive neurodegenerative disorder, affects approximately

1% of the population by the age of 65 years and 4% to 5% of the population by the age of 85 years. Mild cognitive impairment in Parkinson's disease leads to Parkinson's disease dementia (PDD) for which currently there is no drug therapy. The existing treatments for PD were associated with side effects and does not offer complete cure. Hence there is a need of alternative therapy which can prevent or delay the onset of PD with less or no side effects. Vestibular stimulation is known to modulate cognitive processing, enhance learning and spatial memory.

Vestibular dysfunction is present in PD patients. So long term vestibular stimulation may be effective in enhancing cognition by reducing the cognitive, neurodegenerative, neuroinflammatory changes and behavioral deficits observed as predictors of Mild Cognitive Impairment in Parkinson's disease Dementia. In this project, the plan is to administer electric vestibular nerve stimulation to PD patients which might be effective and ideal treatment with minimum or no side effects in the management of Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilled the Hoehn & Yahr Classification of Disability 79,80 stage 1-2
* Ambulate with or without an assistive device for at least 50 feet
* Were able to get up and down from the floor with minimal assistance or less and
* Score of 24 or above on the Folstein Mini-Mental State Exam

Exclusion Criteria:

* Decline in immune function such as pneumonia or systemic infection
* Progressive degenerative disease besides PD
* Spinal fusion or other orthopedic surgery in the past six months
* Mental disease/psychosis such as dementia
* Greater than minimal assistance required for gait and transfers
* Inability to make regular time commitments to the scheduled intervention sessions
* Experience with regular practice of any form of vestibular stimulation within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's disease Rating Scale (UPDRS) | 12 weeks
  The UPDRS has been the most used Parkinsons disease scale. It is a 42 item questionnaire grouped into four subscales. A score of 199 on the UPDRS scale represents the worst (total disability) with a score of zero representing (no disability).

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | 12 weeks
  The 14 item scale is scored by the assessor. Postural stability will be assessed using the Berg balance scale. It assesses the ability of the individual to balance during a series of pre-determined tasks safely. he BBS is a qualitative measure that assesses balance via performing functional activities such as reaching, bending, transferring, and standing that incorporates most components of postural control: sitting and transferring safely between chairs; standing with feet apart, feet together, in single-leg stance, and feet in the tandem Romberg position with eyes open or closed; reaching and stooping down to pick something off the floor. Each item is scored along a 5-point scale, ranging from 0 to 4, each grade with well established criteria. Zero indicates the lowest level of function and 4 the highest level of function. The total score ranges from 0 to 56.
Range of motion (ROM) | 12 weeks
  Range of motion is the available amount of movement of a joint. ROM will be obtained using a universal goniometer and standard protocol.
Muscle Strength | 12 weeks
  Muscle strength will be measured using the Micro FET 2 hand held dynamometer.
Assessment of hand-eye coordination | 12 weeks
  100 pin dexterity test will be performed to assess the speed of coordinated movements. The test requires smooth plastic pad containing fine pierceable100 holes in it and 100 push pins. This set is provided to each participant and is assigned with a task to pin all 100 push pins to the pad. The time required to complete the task will be recorded using a stopwatch. The value will be expressed in seconds.
Assessment of spatial memory | 12 weeks
  20 power point slides presentation will be prepared and projected using a liquid crystal display (LCD) on the screen. Each slide consists of a simple line diagram which is easy to reproduce. Diagrams which could be verbally described like a square, circle, rectangle and pyramid will not included for testing. After showing all the 20 slides, a mathematical problem (e.g., 8-7+3-2+16+12-1+7) will be projected on the screen and asked to solve the problem. Later the participants will be asked to re-call all the 20 slides projected and draw on a paper within a minute. The correct answer are given a score as" 1", and an incorrect answer will be scored as" 0". Different sets of drawings will be used during pre and post assessments
Assessment of verbal memory | 12 weeks
  20 power point slides will be prepared and projected using liquid crystal display (LCD) on the screen. Each slide consists of a three letter word like for example ZOL. After showing all the 20 slides, a mathematical problem (e.g., 9-4+3- 1+22+14-1+3) will be projected on the screen and asked to solve the problem. Later the participants are asked to recall all the 20 slides projected and recollect and present the same on a paper within a minute. The correct answer will be given a score as" 1", and an incorrect answer is scored as" 0". Different sets of drawings will be used during pre and post assessments.
Auditory and visual reaction time | 12 weeks
  Reaction time (RT) apparatus used in the study to record auditory and visual RT was purchased from Anand Agencies, Pune. The RT apparatus presents two auditory (high and low pitch sounds) and two visual stimuli (red and green light).
Estimation of dopamine | 12 weeks
  Dopamine levels will be assessed using General Dopamine (DA) ELISA Kit.
Estimation of Gamma-Aminobutyric Acid (GABA) | 12 weeks
  GABA ELISA Kit will be used to estimate GABA levels
Assessment of quality of life | 12 weeks
  The World Health Organization Quality of Life (WHO-QOL BREF) instrument is a self-administered questionnaire which consists of 26 questions to assess four domains that is physical health, psychological status, social relationships and environment. Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life). The mean score of items within each domain is used to calculate the domain score. Mean scores are then multiplied by 4 in order to make domain scores comparable.
Flexibility | 12 weeks
  Flexibility is the ability of soft tissue structures, such as muscle, tendon, and connective tissue, to elongate through the available range of joint motion. Flexibility measurements will be obtained using a universal goniometer and standard protocol.
Assessment of radiological images | 12 weeks
  MRIs of the cortex, basal ganglia, cerebellum, thalamus, hypothalamus, limbic system and glial cells will be used to assess neurological changes through radiological image data
Assessment of neuronal loss | 12 weeks
  Diameter, area, volume, myelin disruption, gliosis ad=nd connectivity of the neuron will be measured to assess neuronal loss

CONTACTS AND LOCATIONS:
Overall Officials: Sai Sailesh Kumar Goothy, Principal Investigator — RD Gardi Medical College, Ujjain
Locations (1):
- RD Gardi Medical College, Ujjain, Madhya Pradesh, India

REFERENCES:
- [Derived] Kumar Goothy SS, Gawarikar S, Choudhary A, Govind PG, Purohit M, Pathak A, Chouhan RS, Ali Z, Tiwari M, Khanderao MV. Effectiveness of electrical vestibular nerve stimulation on the range of motion in patients with Parkinson's disease. J Basic Clin Physiol Pharmacol. 2022 Oct 10;34(6):791-795. doi: 10.1515/jbcpp-2022-0138. eCollection 2023 Nov 1. PMID 36209355
- [Derived] Kumar Goothy SS, Gawarikar S, Choudhary A, Gajanan Govind P, Purohit M, Pathak A, Chouhan RS, Vijay Khanderao M. Effectiveness of electrical vestibular nerve stimulation as adjunctive therapy to improve the cognitive functions in patients with Parkinson's disease. J Basic Clin Physiol Pharmacol. 2022 Sep 16;34(1):77-82. doi: 10.1515/jbcpp-2022-0066. eCollection 2023 Jan 1. PMID 36103719